CLINICAL TRIAL: NCT05716295
Title: A Phase 1/2, Open-Label, Multicenter Study of MDK-703 as a Monotherapy and in Combination With Other Anti-Cancer Therapies in Patients With Advanced or Metastatic Solid Tumors (ORCHID-1)
Brief Title: A Dose Escalation/Expansion Study of MDK-703 in Patients With Advanced or Metastatic Solid Tumors
Acronym: ORCHID-1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Corporate decision
Sponsor: Medikine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MDK-703-102
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: MDK-703; IL-7; Interleukin 7; Interleukin-7; IL7; oncology; immuno-oncology; immunotherapy; solid tumor; advanced solid tumor; metastatic solid tumor; neoplasms; solid malignancies; pancreatic cancer; PDAC; MSS-CRC; microsatellite stable CRC; microsatellite stable colorectal cancer; prostate cancer; breast cancer; ovarian cancer; immune cold
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Pancreatic Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose escalation followed by dose expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MDK-703 Monotherapy (Experimental): MDK-703 will be administered in sequential ascending doses as a monotherapy until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: MDK-703
- MDK-703 in combination with a checkpoint inhibitor (Experimental): MDK-703 will be administered in sequential ascending doses in combination with a checkpoint inhibitor until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: MDK-703; Drug: Checkpoint Inhibitor, Immune

INTERVENTIONS:
Drug: MDK-703 — MDK-703 will be administered as specified under Arm description.
Drug: Checkpoint Inhibitor, Immune — Checkpoint inhibitor will be administered as specified under Arm description.
  Arms: MDK-703 in combination with a checkpoint inhibitor

SUMMARY:
This is an open-label, dose escalation and dose expansion study of MDK-703 as a monotherapy and in combination with other cancer therapies in adult study participants with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multicenter, dose escalation and dose expansion study evaluating MDK-703 in adult study participants with advanced or metastatic solid tumors. This study will initially commence with dose escalation to evaluate the safety/tolerability of MDK-703 as a monotherapy and in combination with other cancer therapies. Once the monotherapy and/or combination therapy maximum tolerated dose (MTD), optimal biological dose (OBD), and/or recommended dose (RD) has been determined, then dose expansion of MDK-703 may commence in select populations of interest. The study will also evaluate the anti-tumor activity and pharmacokinetic (PK) and pharmacodynamic (PD) profiles of MDK-703 as a monotherapy and in combination with other cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate cardiovascular, hematological, liver, and renal function.
* Prior anti-cancer therapy is allowed as long as any treatment related toxicity is resolved to an appropriate level.
* Females of childbearing potential and men who are not surgically sterile must agree to use medically-accepted method of birth control during the study.
* [Females] Negative serum pregnancy test within 14 days prior to initiating study treatment.
* [Males] Agreement to refrain from donating or banking sperm during the treatment period.

Exclusion Criteria:

* Treated with anti-cancer therapy or an investigational agent within 2 weeks or 5 half-lives prior to first dose, whichever is shorter; or within 4 weeks for immunotherapy.
* Unresolved toxicities from prior systemic therapy greater than NCI CTCAE grade 1 at time of first dose, except alopecia, vitiligo, and grade 2 neuropathy due to prior chemotherapy.
* Radiotherapy within 14 days prior to first dose of study drug.
* Major surgery within 30 days prior to first dose of study drug, or anticipation of major surgery during study treatment.
* Active autoimmune disease requiring systemic treatment within the past 3 months or have a documented history of clinically severe autoimmune disease that requires systemic steroids or immunosuppressive agents.
* Primary central nervous system (CNS) disease or leptomeningeal disease.
* Impaired cardiovascular function or clinically significant cardiovascular disease.
* Uncontrolled diabetes mellitus or other uncontrolled immune-related endocrinopathies.
* Abnormal pulmonary function within the previous 6 months, including history of pneumonitis, active pneumonitis, interstitial lung disease requiring the use of steroids, idiopathic pulmonary fibrosis, active pleural effusion, severe dyspnea at rest or requiring supplementary oxygen therapy.
* History of allogenic, bone marrow, or solid organ transplant.
* History of cerebrovascular events within 6 months prior to first dose.
* Human immunodeficiency virus (HIV) infection or active infection with hepatitis C; uncontrolled hepatitis B infection.
* Clinically significant bleeding within 2 weeks prior to first dose (e.g., gastrointestinal bleeding, intracranial hemorrhage).
* Prior diagnosis of pulmonary embolism within 3 months prior to first dose.
* Known intolerance, hypersensitivity, or contraindication to any components of MDK-703 or checkpoint inhibitors for applicable cohorts.
* History of other malignancy within 5 years prior to first dose, except for patients who are disease-free for >2 years after treatment with curative intent or who have carcinoma in situ which has been excised.
* Any serious medical condition (including pre-existing autoimmune disease or inflammatory disorder), laboratory abnormality, psychiatric condition, or any other significant or unstable concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy or would make the subject inappropriate for the study.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Assessed up to 24 months
  Based on toxicities observed from time of first dose through first cycle of treatment
Maximum tolerated dose (MTD) | Assessed up to 24 months
  Based on toxicities observed
Optimal biological dose (OBD) | Assessed up to 24 months
  Based on toxicities observed
Recommended dose (RD) | Assessed up to 24 months
  Based on toxicities observed
Adverse events (AE) | Assessed up to 24 months
  Incidence and severity of treatment-emergent AEs and serious AEs as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Assessed up to 24 months
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Assessed up to 24 months
  Based on assessment of radiographic imaging per RECIST version 1.1
Time to Response (TTR) | Assessed up to 24 months
  Based on assessment of radiographic imaging per RECIST version 1.1
Disease Control Rate (DCR) | Assessed up to 24 months
  Based on assessment of radiographic imaging per RECIST version 1.1
Progression-Free Survival (PFS) | Assessed up to 24 months
  Based on assessment of radiographic imaging per RECIST version 1.1
Overall Survival (OS) | Assessed up to 24 months
  Based on assessment of radiographic imaging per RECIST version 1.1
Blood concentration of MDK-703 | Assessed up to 24 months
  Blood concentration of MDK-703 at various timepoints
Time to achieve maximum blood concentration | Assessed up to 24 months
  Time to achieve maximum blood concentration of MDK-703

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leveque, MD, Study Director — Chief Medical Officer
Locations (6):
- United States (6):
  - Sarah Cannon Research Institute (Florida Cancer Specialists), Sarasota, Florida
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - NEXT Oncology Austin, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No